CLINICAL TRIAL: NCT01845636
Title: Olfactory Deficits in Mild Cognitive Impairment as a Predictor of Improved Cognition on Donepezil
Brief Title: Olfactory Deficits in MCI as Predictor of Improved Cognition on Donepezil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Davangere P. Devanand, Professor of Clinical Psychiatry and Neurology, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6577; W81XWH-12-0142 (Other Grant/Funding Number: DOD and TATRC)
Record Dates: First submitted 2013-04-26; First posted 2013-05-03 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Olfaction; Donepezil; Alzheimer's Disease; Mild Cognitive Impairment; Memory
MeSH Terms: conditions — Cognitive Dysfunction; Anosmia; Alzheimer Disease | interventions — Donepezil; Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Donepezil Treatment & Atropine Challenge (Experimental): Atropine nasal spray is administered at baseline for the atropine challenge which involves administration of the 40-item University of Pennsylvania Smell Identification Test (UPSIT) immediately before and 45 minutes after atropine administration. Immediately after the atropine challenge, donepezil treatment is started and continues for 52 weeks.
  Interventions: Drug: Donepezil; Drug: Atropine

INTERVENTIONS:
Drug: Donepezil — Donepezil 5mg will be given for 4 weeks and if tolerated, the dose will be increased to 10 mg per day. The dose range of 5 to 10 mg of donepezil per day will be continued for the study duration, and this is the recommended dose for donepezil in the treatment of mild to moderate Alzheimer's disease.
  Other Names: Aricept
Drug: Atropine — A single acute dose of 1 mg of atropine nasal spray is administered to the nostril. The dose chosen reflects clinical doses typically used by Ear, Nose, and Throat (ENT) physicians.
  Other Names: Atropine sulfate ophthalmic solution 1%

SUMMARY:
Odor identification deficits, which are a result of early Alzheimer's Disease (AD) pathology in the olfactory bulb and tract as well as olfactory projection areas in the medial temporal lobe (entorhinal and piriform cortex and hippocampus), lateral and central orbitofrontal cortex and several other regions, occur in AD and strongly predict mild cognitive impairment (MCI) conversion to AD. Our pilot data, along with converging findings in the literature, suggests that odor identification deficits, both incremental change over time and change in response to an anticholinergic challenge, may be clinically simple, relatively inexpensive, predictors of cognitive improvement with acetylcholinesterase inhibitor (ACheI) treatment with potential clinical implications for predicting improvement and monitoring ACheI therapy.

DETAILED DESCRIPTION:
In this clinical trial, the investigators will evaluate, treat and follow a broad sample of 60 adult patients with amnestic MCI at New York State Psychiatric Institute/Columbia University Medical Center. Recruitment will be from clinics and/or advertisements. In the protocol, all 60 amnestic MCI patients will receive baseline memory and olfactory assessments and begin treatment with donepezil. Patients will be followed for a total of 1 year. During this time, patients will be monitored closely by the study physician and will receive memory and olfactory assessments at weeks 8, 26, and 52. In addition, an olfactory challenge test will be done at baseline.

This project will be of value in the selection of patients with mild cognitive impairment for treatment based on the evaluation of olfaction tests to predict response to donepezil and other ACheI. Since mild cognitive impairment is widespread and Alzheimer's disease represents a major public health problem, this study has considerable public purpose and significance.

ELIGIBILITY:
Inclusion Criteria:

* Of either sex, age 55-95 years old
* Patients who meet criteria for amnestic mild cognitive impairment by meeting all of the following:

  (i) subjective memory complaints (ii) Wechsler Memory Scale-R Logical Memory combined Story A + B immediate recall score or combined Story A + B delayed recall score or Free and Cued Selective Reminding Test immediate recall or delayed recall score greater than 1.5 Standard Deviation (SD) below norms or Selective Reminding Test immediate recall or delayed recall score greater than 1.5 SD below norms iii) no functional impairment consistent with dementia
* Folstein Mini Mental State (MMSE) score ≥ 23 out of 30
* Clinical Dementia Rating (CDR) of 0.5 (questionable dementia)
* Availability of informant

Exclusion Criteria:

* Meets Criteria for dementia by Diagnostic and Statistical Manual IV (DSM-IV) criteria or probable Alzheimer's disease
* Meets DSM IV criteria for:

  (i)schizophrenia, schizoaffective disorder, other psychosis, or bipolar I disorder (ii)alcohol or substance dependence or abuse (current or within past 6 months)
* Current untreated major depression or suicidality
* Parkinson's disease, Lewy body disease, multiple sclerosis, central nervous system infection, Huntington's disease, amyotrophic lateral sclerosis, other major neurological disorder.
* Mental Retardation
* Clinical stroke with residual neurological deficits. MRI findings of cerebrovascular disease (small infarcts, lacunes, periventricular disease) in the absence of clinical stroke with residual neurological deficits will not lead to exclusion.
* Patients receiving cholinesterase inhibitors (donepezil, rivastigmine, galantamine) or memantine will be excluded.
* Acute, severe, unstable medical illness. For cancer, patients with active illness or metastases will be excluded, but past history of successfully treated cancer will not lead to exclusion.
* Medical contraindication to donepezil treatment or prior history of intolerability to donepezil treatment.
* Medications with anticholinergic effects that have been shown to adversely impact cognition will not be permitted. Benzodiazepines in lorazepam equivalents greater than or equal to 2 mg daily and narcotics will also not be permitted.
* Exclusion criterion for olfaction: history of anosmia due to any cause (e.g. traumatic or congenital) verified by UPSIT score of <11 out of 40; head trauma with loss of consciousness; nasal sinus disease, current upper respiratory infection; severe allergies to odors; current smoker > 1 pack daily.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davangere Devanand, M.D., Principal Investigator — Columbia University; Gregory Pelton, M.D., Study Director — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donepezil Treatment & Atropine Challenge
Started | 41
Completed | 37
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil Treatment & Atropine Challenge
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37
Selective Reminding Test Total Recall Score [Mean (Standard Deviation); unit: Words] — The Selective Reminding Test (SRT) is a 12-item test of verbal learning and memory. To administer, the researcher will read aloud a list of 12 words. The participant repeats each word aloud to ensure that the word was heard correctly. Immediately following the reading of all 12 words, the participant is asked to recall as many words as possible within the one minute time limit. The participant is then reminded of the words they did not say and asked to recall the list again. This process is repeated for 6 trials. The total immediate recall for all 6 trials is the number that is reported.
  Words | 33.61 (8.15)

OUTCOME MEASURES:

1. Primary Outcome: Selective Reminding Test (SRT)
Description: The Selective Reminding Test (SRT) is a 12-item test of verbal learning and memory. To administer, the researcher will read aloud a list of 12 words. The participant repeats each word aloud to ensure that the word was heard correctly. Immediately following the reading of all 12 words, the participant is asked to recall as many words as possible within the one minute time limit. The participant is then reminded of the words they did not say and asked to recall the list again. This process is repeated for 6 trials. The total immediate recall is the total number of words recalled by the participant from all 6 trials. This is the number that is reported. Lower scores indicate fewer words recalled and a poorer performance.
Time Frame: Week 0, Week 8, Week 26, Week 52
Measure: Mean (Standard Deviation); unit: Words
Arm/Group | Donepezil Treatment & Atropine Challenge
Number analyzed (Participants) | 37
Words
  Week 0 | 33.61 (8.15)
  Week 8 | 36.23 (9.27)
  Week 26 | 36.81 (9.22)
  Week 52 | 37.13 (10.59)

2. Secondary Outcome: Total Number of Errors Measured Using the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Description: The modified Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) is a cognitive battery that assesses learning, memory, language production, language comprehension, constructional praxis, ideational praxis, and orientation. The ADAS-Cog is not a timed test and the participant's score does not depend on how rapidly the test is completed. The ADAS-Cog total score is based on the total number of errors made in the test by the participant. Therefore, a lower total score indicates a higher cognitive performance. The total score ranges from 0 to 95 and is determined by summing the errors from 12 subscales. The total score, indicating number of errors made, is the number that is reported at each timeframe.
Time Frame: Week 0, Week 8, Week 26, Week 52
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Donepezil Treatment & Atropine Challenge
Number analyzed (Participants) | 37
Errors
  Week 0 | 10.67 (4.15)
  Week 8 | 10.27 (3.83)
  Week 26 | 8.80 (3.69)
  Week 52 | 10.09 (4.68)

3. Secondary Outcome: Pfeffer Functional Activities Questionnaire (FAQ)
Description: FAQ is a widely used 10-item instrument that takes 3 minutes to administer and focuses on instrumental, social and cognitive functioning. The assessment is completed by a study informant - typically a caregiver able to report best on the patient's current ability. The instrument assesses the patient's current ability, at the point of testing and through the past month, in these various domains. The total score is described as the cumulative scores of each item, ranging from "0 - No help needed" to "3 - No, unable to do." More impairment is indicated by higher scores. The reported total score range is from 0 (no impairment score) to 30 (maximum impairment score).
Time Frame: Week 0, Week 4, Week 8, Week 26, Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil Treatment & Atropine Challenge
Number analyzed (Participants) | 37
units on a scale
  Week 0 | 3.73 (4.17)
  Week 8 | 4.37 (4.72)
  Week 26 | 4.40 (4.74)
  Week 52 | 5.16 (5.36)

4. Secondary Outcome: Measurement of Everyday Cognition (Ecog)
Description: This instrument has 40 items, takes 20 minutes to administer, and focuses on functional correlates of cognitive deficits. This assessment asks the study informant to rate the participant's ability to perform certain tasks with the domains of Memory, Language, Visual-spatial and Perceptual Abilities, Executive Functioning: Planning, Executive Functioning: Organization, and Executive Functioning: Divided Attention. The informant is asked to compare functioning from 10 years prior to the time of testing. The Everyday Cognition measure uses the sum score of all of the subscales, and the items are reverse coded (i.e., 1= "Better or no change", 2="Questionable/occasionally worse", 3="Consistently a little worse", 4="Consistently much worse"), meaning that lower scores are better. Reported total scores range from 39 (Better or no change) to 156 (Consistently much worse).
Time Frame: Week 0, Week 4, Week 8, Week 26, Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil Treatment & Atropine Challenge
Number analyzed (Participants) | 37
units on a scale
  Week 0 | 60.27 (23.13)
  Week 8 | 62.80 (27.91)
  Week 26 | 63.37 (28.93)
  Week 52 | 65.39 (29.53)

5. Secondary Outcome: Clinician's Interview Based Impression of Change Plus Caregiver Input (CIBIC-plus)
Description: The CIBIC-plus is a well-validated, reliable and widely used measure (range 1-7) of global improvement used in AD and MCI trials. This is a measure of change based on clinician impression.
Time Frame: Week 8, Week 26, Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil Treatment & Atropine Challenge
Number analyzed (Participants) | 37
units on a scale
  Week 8 | 3.43 (0.7)
  Week 26 | 3.31 (0.74)
  Week 52 | 3.13 (1.18)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected beginning at study start in August 2012 and ending at study conclusion in March 2016.
Arm/Group | Donepezil Treatment & Atropine Challenge
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 2/41
Other Adverse Events (participants affected / at risk) | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Treatment & Atropine Challenge (N=41)
Alcohol abuse (Psychiatric disorders) | 1
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes